CLINICAL TRIAL: NCT03555383
Title: Hemostasis Kinetics During Bloodless Liver Transplantation
Brief Title: Individualized Multimodal Hemostasis Evaluation Pyramid (IMHOTEP)
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Janos Fazakas MD, PhD, Research Leader, Semmelweis University
Other Study IDs: Semmelweis University
Record Dates: First submitted 2018-04-24; First posted 2018-06-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Blood Loss, Postoperative; Liver Transplant; Hemostatic Disorder
Keywords: bloodless transplantation; hemostasis reserve capacity; surgery
MeSH Terms: conditions — Postoperative Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coagulation factor levels — The minimal functional hemostasis reserve capacity are defined by triggers as hematocrit: 27%, platelets: 30 G/l, Fibrinogen (FI): 1g/l, FII-FV-FVII-FX: 30%, Antithrombin III: 40%, FXIII: 60% levels. The estimate blood volume methodology is used for to determine the amount of allowable blood loss in volume (ml) that does not require replacement based on current and trigger levels. The individualized pyramid of intervention defined as hemostasis reserve capacity are followed at every studied patient. All measurements and calculations are performed before liver transplantation (T1), at arrival on Intensive Care Unit (T2) and 12-24-48 hours after liver transplantation (T3-4-5).
  Other Names: Calculation of hemostasis reserve capacity

SUMMARY:
This study evaluates the hemostatic changes defined as hemostasis reserve capacity (HRC) in the first perioperative 48 hours of bloodless liver transplanted patients.

DETAILED DESCRIPTION:
The liver transplantation is a common lifesaving procedure with an increased risk of bleeding in end stage liver disease patients. Historically liver transplantation (LT) has been associated with major postoperative blood loss, nevertheless in the last couple of years Massicotte had published increasing number of bloodless liver transplantation (LT) based on acute normovolemic hemodilution, portal pressure reduction and "cell saver" technique and Professor Görlinger many publications underlined the targeted, thromboelastometry guided use of factor concentrates in the background of bloodless liver transplantation. The chronic liver disease is associated with a rebalanced and often pro-coagulant hemostasis, a reduced reserve capacity within the system and a potentially considerable risk for a hemostasis imbalance manifested in microvascular bleeding or thrombosis. The maintenance of blood homeostasis basic condition parallel with the replacement of different coagulation factors according to their reduction order during liver transplantation is highlighted in the Professor Görlinger's pyramid of therapy of coagulopathies, which helps to maintain the hemostasis balance in most of all circumstances. The elevated risk of microvascular bleeding is well circumscribed by low coagulation factor levels in many guidelines, at last in the least European Society of Anesthesia guideline of perioperative bleeding management. However, in certain patients would be unfair to treat standard or viscoelastic tests results according to the guidelines in the absence of clinically manifest coagulopathy. The major objective of this study was to investigate the kinetics of hemostasis reserve capacity (HRC) in the perioperative 48 h of blood products less liver transplantation and absence of surgical and non-surgical bleeding by the implementation of the "Görlinger pyramid methodology" on guidelines directive close or slightly lower hemostasis reserves.

Demographic data of the patients, general: Acute Physiology And Chronic Health Evaluation (APACHE II), Sequential Organ Failure Assessment Score (SOFA) and transplantation specific severity scores Donor Risk Index (DRI), Model For End-Stage Liver Disease (MELD) are recorded along with surgical-, cold- and rewarming ischemia times Cold Ischaemic Time (CIT) Warm Ischaemic Time (WIT) or different organ supports. The hemodynamic parameters as intravascular pressure, volume and flow parameters are followed by transpulmonary volumetric hemodynamic technique (PiCCO2 monitor, Maquet). Standardized laboratory assays and hemostatic tests (Factor I-II-V-VII-X-XIII, AT III) are carried out by Sysmex® CS-2000i, Sysmex® XN-1000 and Siemens® Dimension-RXLMAX systems. Intervention required minimal functional hemostasis reserve capacity are defined by triggers as hematocrit: 27%, platelets: 30 G/l, Fibrinogen (FI): 1g/l, Factor II. (FII.), Factor V (FV.), Factor VII (FVII.), Factor X (FX.): 30%, Antithrombin III: 40%, Factor XIII (FXIII.): 60% levels. The estimate blood volume methodology (EBV, blood volume method) is used for to determine the amount of allowable blood loss in volume (ml) that does not require replacement based on current and trigger levels. According to the algorithm, an individualized pyramid of intervention defined as hemostasis reserve capacity are followed at every studied patient. All measurements and calculations are performed before liver transplantation (T1), at arrival on the Intensive Care Unit (T2) and 12-24-48 h after liver transplantation (T3-4-5). The intraoperative whole blood coagulation is noted by thromboelastographic standard kaolin assay (TEG 5000, Haemonetics®) during hepatectomy, anhepatic phase and end of LT.

Data are analyzed with Statistical Package for the Social Sciences (SPSS, version 20.0, SPSS Inc., Chicago, IL) through descriptive statistics (relative frequency distribution, means and ± Standard Deviation (SD) and inferential statistics (Fischer's exact test and r-ANOVA). In all tests, an a priori alpha error p-value of less than 0.05 and confidence intervals (CI) of 95% are considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All bloodless liver transplanted patients in Semmelweis University Department of Transplantation and Surgery will be included in the study

Exclusion Criteria:

* Patients with:

Required Red Blood Cells (RBC), Fresh Frozen Plasma (FFP) or platelets replacement in the perioperative first 48 hours, pediatric patients (age < 18 years) and acut liver failure patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent bloodless liver transplantation in Semmelweis University Department of Transplantation and Surgery
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change of coagulation factor levels and hemostasis reserve capacity during bloodless liver transplantation from baseline till the second postoperative day | Participants will be followed preoperatively, postoperative 0,12, 24, 48. hours after liver transplantation
  Based on coagulation factors measurements the allowable blood loss is calculated and defined as hemostasis reserve capacity till compulsory coagulation factor or blood products replacement is needed to avoid coagulopathic bleeding in the perioperative phase of liver transplantation. The changes of the measured coagulation factors and the hemostasis reserve capacity is counted at the different meaning points: baseline-before liver transplantation (T1), after successful liver transplantation at arrival on intensive care unit-ICU (T2) and postoperatively according to the graft function: 12 hours after liver transplantation (T3), 24 hours after liver transplantation (T4), 48 hours after liver transplantation (T5).

SECONDARY OUTCOMES:
Length of Intensive Care Unit stay | An expected average of 3 days
  Participants will be followed for the duration of Intensive Care Unit stay
Length of hospital stay | An expected average of 2 weeks
  Participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baron DM, Metnitz PG, Fellinger T, Metnitz B, Rhodes A, Kozek-Langenecker SA. Evaluation of clinical practice in perioperative patient blood management. Br J Anaesth. 2016 Nov;117(5):610-616. doi: 10.1093/bja/aew308. PMID 27799175
- [Background] Bidlingmaier C, Olivieri M, Hutker S, Dietl S, Kurnik K. Perioperative management of hemostasis in children and adolescents. Blood Cells Mol Dis. 2017 Sep;67:91-95. doi: 10.1016/j.bcmd.2017.01.009. Epub 2017 Jan 16. PMID 28130047
- [Background] Gibon E, Courpied JP, Hamadouche M. Total joint replacement and blood loss: what is the best equation? Int Orthop. 2013 Apr;37(4):735-9. doi: 10.1007/s00264-013-1801-0. Epub 2013 Feb 6. PMID 23385607
- [Background] Goel R, Cushing MM, Tobian AA. Pediatric Patient Blood Management Programs: Not Just Transfusing Little Adults. Transfus Med Rev. 2016 Oct;30(4):235-41. doi: 10.1016/j.tmrv.2016.07.004. Epub 2016 Aug 1. PMID 27559005
- [Background] Gorlinger K. [Coagulation management during liver transplantation]. Hamostaseologie. 2006 Aug;26(3 Suppl 1):S64-76. German. PMID 16953295
- [Background] Kahvecioglu D, Erdeve O, Alan S, Cakir U, Yildiz D, Atasay B, Arsan S. The impact of evaluating platelet transfusion need by platelet mass index on reducing the unnecessary transfusions in newborns. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1787-9. doi: 10.3109/14767058.2013.879708. Epub 2014 Feb 3. PMID 24397345
- [Background] Keir AK, Stanworth SJ. Neonatal Plasma Transfusion: An Evidence-Based Review. Transfus Med Rev. 2016 Oct;30(4):174-82. doi: 10.1016/j.tmrv.2016.07.001. Epub 2016 Jul 9. PMID 27473518
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785
- [Background] Lang H, Mouracade P, Gimel P, Bernhard JC, Pignot G, Zini L, Crepel M, Rigaud J, Salomon L, Bellec L, Vaessen C, Roupret M, Jung JL, Mourey E, Martin X, Bigot P, Bruyere F, Berger J, Ansieau JP, Salome F, Hubert J, Pfister C, Trifard F, Gigante M, Baumert H, Mejean A, Patard JJ. National prospective study on the use of local haemostatic agents during partial nephrectomy. BJU Int. 2014 May;113(5b):E56-61. doi: 10.1111/bju.12397. Epub 2013 Oct 31. PMID 24053412
- [Background] Massicotte L, Denault AY, Thibeault L, Hevesi Z, Nozza A, Roy A. Relationship between conventional coagulation tests and bleeding for 600 consecutive liver transplantations. Transplantation. 2014 Jul 27;98(2):e13-5. doi: 10.1097/TP.0000000000000253. No abstract available. PMID 25022237